CLINICAL TRIAL: NCT00204477
Title: Soybean Diet and Breast Density
Brief Title: Soy Protein and Breast Cancer Risk Reduction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02-422; Army's HSRRB log no. A-10926 (Other: USA MRMC Human Research Protection Office (HRPO)); UTMB GCRC 533 (Other: UTMB ITSCRC); DAMD17-01-1-0417 (Other Grant/Funding Number: USA MRMC); M01RR000073 (NIH); 1UL1RR029876-01 (NIH)
Record Dates: First submitted 2005-09-09; First posted 2005-09-20 (Estimated); Results first posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: soy diet; breast cancer; ovarian hormones; breast density; prevention
MeSH Terms: conditions — Breast Neoplasms | interventions — Soy Milk; Milk

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled, 2 parallel groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research pharmacist dispensed blinded assigned sachets according to a pre-generated randomization list. Pharmacists were blinded to all other aspects of the research protocols.
  Subjects, investigators, research staff, and statisticians were all blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soy milk (Active Comparator): Subjects will consume two soy milk drinks from the content of 2 sachets (40 g isoflavone-free soy protein and 600 mg calcium) in place of a small meal, five days per week. Each sachet will contain 20 g soy protein and 300 mg calcium. Content of sachets will be mixed with ~1.6 liter of water for ingestion.
  Interventions: Dietary Supplement: soy milk
- Cow's milk (Placebo Comparator): Subjects will consume two cow's milk drinks from the content of 2 sachets (40 g cow's milk protein, casein, and 600 mg calcium) in place of a small meal, five days per week. Each sachet will contain 20 g cow's milk protein and 300 mg calcium. Content of sachets will be mixed with ~1.6 liter of water for ingestion. Casein is free of ovarian hormones.
  Interventions: Dietary Supplement: cow's milk

INTERVENTIONS:
Dietary Supplement: soy milk — Each drink contained soy protein, fat, and carbohydrates calcium and phosphorous to give a total energy of 177.8 kcal. Subjects took two drinks per day.
  Other Names: Not applicable, research product
  Arms: Soy milk
Dietary Supplement: cow's milk — Each drink contained casein, fat, carbohydrates, calcium and phosphorous to give a total energy of 178.6 kcal. Subjects took two drinks per day.
  Other Names: Not applicable, research product
  Arms: Cow's milk

SUMMARY:
Soy consumption has been associated with reduced risk for developing breast cancer. Ovarian hormones and breast density are considered breast cancer risk markers. We propose to test the hypothesis that consumption of soy protein reduces ovarian steroid hormones and results in a corresponding reduction in breast density comparing to casein protein.

DETAILED DESCRIPTION:
The aims will be tested by conducting a randomized, double-blind study, with two arms and 100 women in each arm. Premenopausal women will be recruited and randomly allocated to take one of two different dietary supplements daily for 2 years. The two test diets soy protein drink and caseinate protein drink. Multiple blood, urine, and breast fluid samples will be obtained before and during the dietary intervention period and analyzed for ovarian hormones. At baseline and after the intervention period, breast density, and bone density will be assessed by radiological techniques at baseline and 1 yr and 2 yr after protein drink supplementation. The efficacy of the dietary intervention will be determined by comparing mean changes of ovarian steroids, and density of the breast and bone tissues over the 2 year dietary intervention period in the two diet groups with adjustment for baseline values and individual patient characteristics of interest. We predict that 2 years of soya dietary supplements will reduce breast density, which will be explained by individual hormonal changes.

ELIGIBILITY:
Inclusion Criteria:

* healthy premenopausal women
* 30 to 40 years old
* normal mammograms
* regular menstrual cycles

Exclusion Criteria:

* abnormal mammograms
* first degree relatives with breast cancer
* pregnant or lactating
* peri- or post-menopause
* breast augmentation, reduction, and lifting
* on oral contraceptive medications or exogenous hormones
* medically prescribed diets
* allergic reaction to soy or cow's milk

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only females with regular monthly menstrual cycles, not expecting to become pregnancy, not breast feeding, and not on contraceptives
Enrollment: 321 (Actual)
Dates: Start 2002-04 (Actual); Primary Completion 2011-07-22 (Actual); Study Completion 2023-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee-Jane W Lu, Ph.D., Principal Investigator — The University of Texas Medical Branch, Galveston, TX 77555
Locations (1):
- General Clinical Research Center, The University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Will not share as this required financial resources.

REFERENCES:
- [Derived] Lu LJ, Nishino TK, Johnson RF, Nayeem F, Brunder DG, Ju H, Leonard MH, Grady JJ, Khamapirad T. Comparison of breast tissue measurements using magnetic resonance imaging, digital mammography and a mathematical algorithm. Phys Med Biol. 2012 Nov 7;57(21):6903-27. doi: 10.1088/0031-9155/57/21/6903. Epub 2012 Oct 9. PMID 23044556
- [Derived] Nayeem F, Anderson KE, Nagamani M, Grady JJ, Lu LJ. Alkaline phosphatase and percentage body fat predict circulating C-reactive protein in premenopausal women. Biomarkers. 2010 Dec;15(8):663-70. doi: 10.3109/1354750X.2010.509811. Epub 2010 Sep 29. PMID 20874659

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Soy Milk | Cow's Milk
Started | 161 | 160
Completed | 161 | 160
Not Completed | 0 | 0
Period: One Year After Diet
Arm/Group | Soy Milk | Cow's Milk
Started (Picked up the diet) | 128 | 125
Completed (Complete 1 year of diet) | 86 | 87
Not Completed | 42 | 38
Not completed — Did not complete 1 year of diet | 42 | 38
Period: Two Years After Diet
Arm/Group | Soy Milk | Cow's Milk
Started (Complete full 2nd year of diet.) | 55 | 62
Completed | 39 | 49
Not Completed | 16 | 13
Not completed — Did not complete the 2nd year of diet | 16 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Soy Milk | Cow's Milk | Total
Number analyzed (Participants) | 161 | 160 | 321
Age, Customized [Number; unit: years]
  Ages from 29 to 41 | 161 | 0 | 161
  Agesfrom 30 to 41 | 0 | 160 | 160
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 160 | 321
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan | 1 | 0 | 1
  Asian | 2 | 3 | 5
  Black/African American | 21 | 18 | 39
  Hispanic or Latino | 57 | 71 | 128
  Other (>2 races) | 3 | 2 | 5
  Caucasian | 77 | 66 | 143
Region of Enrollment [Number; unit: participants]
  United States | 161 | 160 | 321

OUTCOME MEASURES:

1. Primary Outcome: Mammographic Density (Baseline)
Description: Breast images were acquired by digital mammography. Fibroglandular tissue were segmented from fatty breast tissue. The total breast area is the sum of the fibroglandular tissue area and fatty breast tissue area. Mammographic density (breast density) is the percentage of fibroglandular tissue in the total breast.
Time Frame: Baseline
Population: 4 participants images in the cow's milk and 3 images in soy milk were either missing or corrupt.
Measure: Mean (Standard Deviation); unit: percentage of glandular tissue in breast
Arm/Group | Soy Milk | Cow's Milk
Number analyzed (Participants) | 157 | 157
percentage of glandular tissue in breast | 29.21 (11.44) | 28.24 (11.77)

2. Primary Outcome: Mammographic Density (1 Year)
Description: as for outcome 1
Time Frame: 1 Year
Population: Participants completed one year of diet.
Measure: Mean (Standard Deviation); unit: percentage of glandular tissue in breast
Arm/Group | Soy Milk | Cow's Milk
Number analyzed (Participants) | 86 | 87
percentage of glandular tissue in breast | 29.37 (12.78) | 28.01 (11.56)

3. Primary Outcome: Mammographic Density (2 Years)
Description: as for outcome 1
Time Frame: 2 years
Population: Participants completed 2 years of study. 1 image missing from the cow's milk group due to it was corrupt.
Measure: Mean (Standard Deviation); unit: percentage of glandular tissue in breast
Arm/Group | Soy Milk | Cow's Milk
Number analyzed (Participants) | 39 | 48
percentage of glandular tissue in breast | 30.75 (13.26) | 29.06 (11.80)

4. Primary Outcome: Breast Tissue Composition Measured by MRI
Description: Breast images acquired by breast magnetic resonance imaging (MRI). The amount of fatty breast tissue,(cc), glandular breast tissue(cc ), total breast (cc), and percentage of glandular tissue in total breast (%) were estimated.
Time Frame: Baseline
Population: 4 participants images in the cow's milk and 14 images in soy milk were either missing or corrupt.
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Soy Milk | Cow's Milk
Number analyzed (Participants) | 147 | 156
cc
  Fatty Breast Tissue, cc | 589.9 (333.5) | 628.1 (373.4)
  Glandular Breast Tissue, cc | 153.4 (84.48) | 156.7 (88.75)
  Total Breast, cc | 743.3 (350.9) | 784.9 (400.8)

5. Primary Outcome: Breast Tissue Composition Measured by MRI
Description: as for outcome 4
Time Frame: 1 Year
Population: Participants completed year 1.
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Soy Milk | Cow's Milk
Number analyzed (Participants) | 86 | 86
cc
  Fatty Breast Tissue, cc | 587.4 (341.8) | 626.1 (358.9)
  Glandular Breast Tissue, cc | 159.3 (89.72) | 156.7 (83.06)
  Total Breast, cc | 746.7 (358.8) | 782.8 (387.5)

6. Primary Outcome: Breast Tissue Composition Measured by MRI
Description: as for outcome 4
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Soy Milk | Cow's Milk
Number analyzed (Participants) | 39 | 49
cc
  Fatty Breast Tissue, cc | 629.9 (406.5) | 615.5 (395.9)
  Glandular Breast Tissue, cc | 173.8 (104.5) | 152.7 (87.44)
  Total Breast, cc | 803.7 (420.8) | 768.2 (426.4)

7. Other Pre Specified Outcome: Blood Will be Measured for Standard Clinical Chemistries
Description: Serum will be measured for for blood chemistries , 4 times at baseline, and thereafter at 3-monthly interval for up to 2 years of protein drink supplementation
Time Frame: 4 measurements at baseline and once every three months after protein drink supplements for up to 2 years.
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Progesterone (ng/ml)
Description: Serum will be measured for progesterone (ng/ml), 4 times at baseline, and thereafter at 3-monthly interval for up to 2 years of protein drink supplementation
Time Frame: 4 measurements at baseline and once every three months after protein drink supplements for up to 2 years.
Reporting Status: Not Posted

9. Primary Outcome: Percentage of Grandular Tissue in Total Breast Measured by MRI
Description: as for outcome 4
Time Frame: Baseline
Population: 4 participants images in the cow's milk and 14 images in soy milk were either missing or corrupt.
Measure: Mean (Standard Deviation); unit: % of glandular tissue in total breast
Arm/Group | Soy Milk | Cow's Milk
Number analyzed (Participants) | 147 | 156
% of glandular tissue in total breast | 24.27 (13.64) | 24.09 (15.83)

10. Primary Outcome: Percentage of Grandular Tissue in Total Breast Measured by MRI
Description: as for outcome 4
Time Frame: 1 Year
Population: Participants completed year 1.
Measure: Mean (Standard Deviation); unit: % of glandular tissue in total breast
Arm/Group | Soy Milk | Cow's Milk
Number analyzed (Participants) | 86 | 86
% of glandular tissue in total breast | 25.017 (14.48) | 24.20 (15.82)

11. Primary Outcome: Percentage of Grandular Tissue in Total Breast Measured by MRI
Description: as for outcome 4
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: % of glandular tissue in total breast
Arm/Group | Soy Milk | Cow's Milk
Number analyzed (Participants) | 39 | 49
% of glandular tissue in total breast | 26.39 (15.52) | 24.25 (15.89)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Soy Milk | Cow's Milk
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/160
Serious Adverse Events (participants affected / at risk) | 0/161 | 0/160
Other Adverse Events (participants affected / at risk) | 28/161 | 21/160
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Soy Milk (N=161) | Cow's Milk (N=160)
accident (Musculoskeletal and connective tissue disorders) | 1 | 0
appendectomy (Gastrointestinal disorders) | 1 | 0
hypertension (Cardiac disorders) | 1 | 0
blurred vision (Eye disorders) | 1 | 0
optic migraines (Nervous system disorders) | 1 | 0
Heavy bleeding and uterine polyp (Reproductive system and breast disorders) | 1 | 0
cholecystectomy (Surgical and medical procedures) | 2 | 0
accident (Musculoskeletal and connective tissue disorders) | 1 | 0 — broken left wrist
pregnancy (Pregnancy, puerperium and perinatal conditions) | 5 | 4
urinary tract infection and kidney stones (Renal and urinary disorders) | 1 | 0
fever, abdominal pain, leucopenia of unknown etiology (General disorders) | 1 | 0
strep throat (Infections and infestations) | 1 | 1
enlarged uterus and large fibroids (Reproductive system and breast disorders) | 1 | 0
idiopathic thrombocytopanic purpura (Blood and lymphatic system disorders) | 1 | 0
mild stroke (Nervous system disorders) | 1 | 0
adenopathy in both axilla (Infections and infestations) | 1 | 0
ovariectomy (1) and follipian tube removed (Surgical and medical procedures) | 0 | 1
fever, earache, and hearing loss in left ear (Infections and infestations) | 0 | 1
bladder infection (Infections and infestations) | 0 | 1
accident, fall, rib broke, ankle sprained (Musculoskeletal and connective tissue disorders) | 0 | 1
right breast lump (Skin and subcutaneous tissue disorders) | 0 | 1
recurrent endometriosis, surgery (Surgical and medical procedures) | 0 | 1
tosillitis and UTI (Infections and infestations) | 0 | 1
sprain/fracture wrist (Musculoskeletal and connective tissue disorders) | 0 | 1
blood nipple, one (Blood and lymphatic system disorders) | 0 | 1
laparoscopic lap band elective surgery (Surgical and medical procedures) | 0 | 1
allergic reaction (Immune system disorders) | 0 | 1
fibroid, irregular bleeding (Reproductive system and breast disorders) | 0 | 1
goiter surgery (Surgical and medical procedures) | 0 | 1
tattoos removal (General disorders) | 0 | 1
fibroadnoma of right breast (Reproductive system and breast disorders) | 0 | 1
uterus, laproscopy, D&C (Reproductive system and breast disorders) | 1 | 0
cervix, polyp, bacterial vaginosis (Reproductive system and breast disorders) | 1 | 0
leucopenia, fever, abdominal pain (Infections and infestations) | 1 | 0
accident (General disorders) | 1 | 0 — car accident
pre existing abnormal pap (Reproductive system and breast disorders) | 1 | 0
accident (Musculoskeletal and connective tissue disorders) | 1 | 0 — bicycle accident
leiomyomata (Reproductive system and breast disorders) | 1 | 0
Breast calcification, increase (Reproductive system and breast disorders) | 0 | 1
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No